CLINICAL TRIAL: NCT01886261
Title: Validation of Objective Measures of Place-Based Physical Activity
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Other Study IDs: 111274/ 121378; R01CA167693 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-06-25 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Physical Activity
Keywords: validation; physical activity; place-based interventions; construct validity; divergent validity; usability; gps; PALMS
MeSH Terms: conditions — Motor Activity; Gray Platelet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Usability of the PALMS system, validity of the PALMS system and added value to an existing cohort study.

Hypothesis: Addition of GPS device and use of PALMS system will allow researchers to better examine place-based interventions.

DETAILED DESCRIPTION:
The Personal Activity Location Measurement System (PALMS) researchers at UCSD have created a web-based processing system for location (GPS) and physical activity (accelerometer) data. We will collect data on a pilot sample of 40 Hispanic persons to a) test the validity of PALMS assessments of transportation modes, and activity in different locations against an objective record of activities derived from images collected by Vicon Revue; b) compare PALMS assessments of transportation modes and activity locations to other self-report measures and interview measures; c) assess the construct validity of PALMS-based activity assessment.

We will be assessing the usability of PALMS in a research staff with no previous experience of using the PALMS system. We will be assessing the added value of using PALMS to examine a place-based intervention in an existing cohort study.

ELIGIBILITY:
Validation Study

Inclusion Criteria:

* Adults (18+ years old)
* Self-identify as Hispanic/Latino(a)
* Have a variety of primary transportation modes
* Have a variety of physical activity levels both occupational and leisure
* Commute different distances to the location

Exclusion Criteria:

* Illness that prevents normal activities
* Inability to ambulate
* Unable to wear the devices for up to 7 days
* Unable to complete two phone interviews in English or Spanish
* Unable to complete a written survey in English or Spanish

Usability Testing:

Research staff members of the SDSU Fe en Accion research study.

Added Value Cohort: Fe en Accion

Inclusion Criteria (Participants of the cohort):

* Attend church weekly
* Age: 18 - 65 years old
* Must live in San Diego County
* Live within 4 miles of their church
* engage in less than 150 minutes of leisure time moderate and vigorous physical activity
* Latina woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Validation Study: We will be recruiting 40 primarily Spanish speaking, adults from various community locations throughout San Diego County.
  Usability Testing:
  Recruiting research staff member from the SDSU Fe en Accion research study to participate in usability testing.
  Added Value Cohort: Fe en Accion Participants of the Fe en Accion cohort.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Construct Validity | 7 days
  Construct validity assesses the theoretical relationship of a measure (and resulting variables) with other variables. The multitrait-multimethod matrix (MTMM) is a procedure first developed by Campbell and Fiske to asses construct validity by creating a fully crossed method-by-measure matrix of associations among multiple constructs and multiple measurement methods. The resulting matrix of correlation coefficients gives a pattern of associations that informs the validity evidence of the measure and construct. We will use the following measures in the multitrait multimethod matrix: Neighborhood Physical Activity Questionnaire, the American Timeuse Survey, and PALMS based physical activity in location estimates.
Usability | 1 day
  Direct observation of research staff with no experience using the PALMS system.
Added Value | baseline and 1 year
  We will be assessing GPS tracks in participants in the Fe en Accion cohort to determine the effectiveness of the place-based intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States